## Postural and Muscle Fatigue Analysis of Endodontic Residents

Informed consent form February 2024

## Informed Consent Form

| Study Title: Risk for the development of musculoskeletal disorders in students of the Master's |
|---|
| Degree in Advanced Endodontics, Universidad Europea de Madrid. |

Sponsor: European University of Madrid

Investigators: Antonio Conde (UEM), Gaizka Loroño (UEM), Ruth Pérez (UEM), Roberto Estévez (UEM), Victor Díaz-Flores García (UEM), Juan Carlos Ortiz-Hugues (Panamá), Carlos G. Adorno (UNA, Paraguay)

| Center: European University of Madrid. | | |
|----------------------------------------|----|-------|
| In Madrid, at | of | of 20 |

Dear patient: Your participation is requested in this research project, whose main objective is to determine whether the postures adopted by students of the Master's Degree in Advanced Endodontics during clinical care constitute a risk for the development of temporomuscular disorders (TMD).

During the performance of root canal treatment on an upper or lower molar in the patient, the posture adopted by the student during a part of the treatment will be recorded from 3 different angles (2 lateral and one frontal).

The recording will not interfere with the treatment, which will follow the standard protocols of the clinic. The personal information collected for the study will only be on which tooth the root canal treatment was performed.

No other patient identifiable information will be collected. In case your face appears in the recordings, it will be pixelated or covered from the videos or images that will be used for scientific dissemination in conferences, classrooms and scientific articles, among others.

You will be asked for your consent to participate in the study as a patient of the Advanced Endodontics Master's student. Your participation is completely voluntary, and if you decide not to participate you will receive all the dental care you require and your relationship with the dental team will not be affected.

You must give your informed consent in writing, signing this document so that the tooth to be treated according to the indication is used in the study.

## **Informed Consent**

Title of the study: Risk for the development of musculoskeletal disorders in students of the Master of Advanced Endodontics, Universidad Europea de Madrid.

Sponsor: European University of Madrid Investigators: Antonio Conde (UEM), Gaizka Loroño (UEM), Ruth Pérez (UEM), Roberto Estevez (UEM), Victor Díaz-Flores García (UEM), Juan Carlos Ortiz-Hugues (Panamá), Carlos G. Adorno (UNA, Paraguay).

Center: European University of Madrid.

| Mr./Ms | | , aged <sub>.</sub> | , with ID |
|-------------|----------------|---------------------|-----------|
| card number | and address at | | · |

I have received a satisfactory explanation of the study procedure, its purpose, risks, benefits and alternatives. I have been satisfied with the information received, I have understood it, all

| my doubts have been answ<br>consent for the proposed p<br>the only obligation to infor | procedure and | I know my ri | ight to with | ndraw it when | ever I wish, with |
|---|---|---|---|---|---|
| In Madrid, on the day | of | of | 20 | _· | |
| Signature and ID card num | ber of the inve | stigator Sign | ature and | ID card numbe | er of the patient |
| *In cases of minors between<br>the minor (with the inform<br>corresponding to an adoles<br>of minors under 12 years of | native text adapt<br>scent) and one<br>of age, only the | oted to the use for the legal repres | inderstand<br>I represent<br>entative si | ing and treatn<br>ative of that n<br>gns the conse | nent<br>ninor. In the case |
| both cases varies in the firs | | | | | |
| Mr./Msrepresentative of Mr./Ms. | | , aged,<br>, | _, with ID (<br>aged | card<br>, with ID card <sub>.</sub> | , legal<br>, |
| Signature and ID card num | har of the nati | ont's logal re | nrocontati | V0 | |

Signature and ID card number of the patient's legal representative